CLINICAL TRIAL: NCT02748226
Title: Korean Vascular Intervention Society Multicenter Registry Study on Outcomes of Endovascular Therapy in Lower Limb Artery Diseases (K-VIS ELLA): (A Retrospective & Prospective Observational Study)
Status: Recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2013-0463
Record Dates: First submitted 2016-04-05; First posted 2016-04-22 (Estimated); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Peripheral Arterial Disease(PAD)
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective cohort: This cohort retrospectively enrolls patients with lower extremity artery disease who underwent endovascular treatment from January 2006 to the date of approval by IRB in the participating hospitals.
  Interventions: Procedure: endovascular treatment
- Prospective cohort: This cohort prospectively enrolls patients with lower extremity artery disease who undergo endovascular treatment from the date of approval by IRB to July, 2018 in the participating hospitals.
  Interventions: Procedure: endovascular treatment

INTERVENTIONS:
Procedure: endovascular treatment — endovascular treatment

SUMMARY:
1. Study design: multicenter retrospective and prospective observational study
2. Study Cohort :

   1. Retrospective cohort: This cohort retrospectively enrolls patients with lower extremity artery disease who underwent endovascular treatment from January 2006 to the date of approval by IRB in the participating hospitals. Informed consent was waived by IRB.
   2. Prospective cohort: This cohort prospectively enrolls patients with lower extremity artery disease who undergo endovascular treatment from the date of approval by IRB to July, 2018 in the participating hospitals. Informed consent will be obtained prior to enrollment.
3. Baseline clinical and lesion characteristics, procedural and post-procedural data, clinical outcomes, hemodynamic, and imaging follow-up data are investigated. Primary patency and target lesion revascularization rates of the total cohort and patient subgroups are evaluated. Risk factors of restenosis and target lesion revascularization are determined.

DETAILED DESCRIPTION:
This is an observational study. The study includes patients who underwent endovascular treatments for lower extremity artery diseases and investigates immediate and late outcomes of the treatments. The investigator does not assign any specific interventions.

ELIGIBILITY:
Inclusion Criteria:

* Retrospective data Patients who underwent or attempted endovascular treatment for symptomatic peripheral artery disease from January 2006 until IRB approval date
* Prospective data

  1. Age 20 years of older
  2. Patients in the treatment or trying about symptomatic peripheral artery disease from IRB approval date
  3. Symptomatic peripheral artery disease:

     * Intermittent claudication (Rutherford category 1 to 3)
     * Critical limb ischemia (Rutherford category 4 to 6)

Exclusion Criteria:

1. Pregnant women or women with potential childbearing
2. Moderate Alzheimer's disease, mental illness or neurological disease of more than those who can not understand the purpose of this clinical trials and Methods
3. Life expectancy <1 year due to comorbidity

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lower extremity artery disease
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2013-09-30 (Actual); Primary Completion 2032-07-31 (Estimated); Study Completion 2032-07-31 (Estimated)

PRIMARY OUTCOMES:
Primary patency | 12 months
  Primary patency is defined as freedom from more than 50% restenosis based on CT angiography, duplex ultrasound or catheter-based angiography or from clinically-driven target lesion revascularization.

SECONDARY OUTCOMES:
Target lesion revascularization (TLR) | 12 months
  Any re-intervention within the target lesion due to symptom aggravation or drop of ankle brachial index (ABI) >0.15 when compared to post procedure baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim YH, Her AY, Ko YG, Ahn CM, Lee SJ, Hong MK, Yu CW, Lee JH, Lee SW, Youn YJ, Yoon CH, Rha SW, Min PK, Choi SH, Chae IH, Choi D; K-VIS ELLA Investigators. Drug-coated balloon versus drug-eluting stent for femoropopliteal total occlusions: intraluminal versus subintimal approaches. Sci Rep. 2024 Sep 11;14(1):21173. doi: 10.1038/s41598-024-71745-0. PMID 39256427
- [Derived] Roh JW, Shin S, Ko YG, Son NH, Ahn CM, Min PK, Lee JH, Yoon CH, Yu CW, Lee SW, Lee SR, Choi SH, Chae IH, Choi D. Long-Term Clinical Outcomes of Iliac Artery Endovascular Therapy in the Korean Vascular Intervention Society Endovascular Therapy in Lower Limb Artery Diseases (K-VIS ELLA) Registry. Korean Circ J. 2022 Jul;52(7):529-540. doi: 10.4070/kcj.2021.0390. Epub 2022 Mar 28. PMID 35491481
- [Derived] Cha JJ, Kim JY, Kim H, Ko YG, Choi D, Lee JH, Yoon CH, Chae IH, Yu CW, Lee SW, Lee SR, Choi SH, Koh YS, Min PK; K-VIS (Korean Vascular Intervention Society) investigators. Long-term Clinical Outcomes and Prognostic Factors After Endovascular Treatment in Patients With Chronic Limb Threatening Ischemia. Korean Circ J. 2022 Jun;52(6):429-440. doi: 10.4070/kcj.2021.0342. Epub 2022 Feb 10. PMID 35257522
- [Derived] Lim C, Won H, Ko YG, Lee SJ, Ahn CM, Min PK, Lee JH, Yoon CH, Yu CW, Lee SW, Lee SR, Choi SH, Chae IH, Choi D; K-VIS Investigators. Association between Body Mass Index and Clinical Outcomes of Peripheral Artery Disease after Endovascular Therapy: Data from K-VIS ELLA Registry. Korean Circ J. 2021 Aug;51(8):696-707. doi: 10.4070/kcj.2021.0040. PMID 34327883
- [Derived] Kim J, Park TK, Choi KH, Choi D, Ko YG, Lee JH, Yoon CH, Chae IH, Yu CW, Min PK, Lee SW, Lee SR, Koh YS, Choi SH; Korean Vascular Intervention Society (K-VIS) Endovascular therapy in Lower Limb Artery diseases (ELLA) Registry Investigators. Different association between renal dysfunction and clinical outcomes according to the presence of diabetes in patients undergoing endovascular treatment for peripheral artery disease. J Vasc Surg. 2020 Jan;71(1):132-140.e1. doi: 10.1016/j.jvs.2019.03.071. Epub 2019 Jul 5. PMID 31285068